CLINICAL TRIAL: NCT00901654
Title: A Phase I, Single Center, Double-Blind, Placebo-controlled Dose Finding Clinical Study to Evaluate the Safety and Immunogenicity of the Live Attenuated, Oral Vaccine ACE527
Brief Title: ACE527 Safety and Immunogenicity Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TD Vaccines A/S (Industry)
Collaborators: Pierrel Research USA, Inc. (Industry); Johns Hopkins University (Other)
Responsible Party: Ingelise Saunders/CEO, TD Vaccines A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACE527-101
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Enterotoxigenic E. Coli (ETEC) Infection
Keywords: Vaccination; Diarrhea; Traveler's Diarrhea; ETEC; Enterotoxigenic E. coli
MeSH Terms: conditions — Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE527 (Experimental)
  Interventions: Biological: ACE527 vaccine
- Placebo comparator (Placebo Comparator)
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: ACE527 vaccine — First cohort: Two doses, each of 3x10^9 cfu of each strain (9x10^9 cfu total per dose) administered on Days 0 and Day 21 (out-patient).
  Second cohort: Two doses, each of 3x10^10 cfu of each strain (9x10^10 cfu total per dose) administered on Days 0 and Day 21
  Arms: ACE527
Biological: Placebo vaccine — First and second cohort: The placebo vaccine will be administered at Days 0 and Days 21.
  Arms: Placebo comparator

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to ACE527.

DETAILED DESCRIPTION:
The study is a phase I, single center, double-blind, placebo-controlled dose finding clinical study to evaluate the safety, tolerability and immunogenicity of the live attenuated, oral vaccine ACE527. The study is designed to evaluate 2 doses of the ACE527 in 2 cohorts. Each cohort will consist of approximately 18 subjects (healthy subjects), approximately 12 of them receiving ACE527 and approximately 6 receiving placebo.

Within a cohort, the second dose will only be given if safety and tolerability of the first dose is acceptable. This assessment will be based on evaluation of data up until Day 7 by the Independent Safety Committee (ISC) as per written guidance. The first dose of each cohort will be administered during an inpatient stay. Escalation to the next dose level will be dependent on an acceptable safety profile of the first dose at the previous dose level, based on evaluation of safety data by an Independent Safety Committee (ISC). The decision to administer the second dose at the higher level will also require review of the safety and tolerability of the second dose at the lower level.

The second dose will be administered at the outpatient clinic and the subjects will be observed for at least 60 minutes after vaccination prior to discharge from unit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥18 and ≤50 years.
* General good health, without clinically significant medical illness, physical examination findings or laboratory abnormalities, as determined by the Principal Investigator (PI) or PI in consultation with the medical monitor (MM) and sponsor.
* Negative serum pregnancy test at screening and a negative urine pregnancy test before immunization for female subjects of childbearing potential. Females of childbearing potential must not be breastfeeding and must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female subjects unable to bear children (e.g. tubal ligation or hysterectomy) must have negative pregnancy tests.

Exclusion Criteria:

* Working as a food handler, in child-care or as a healthcare worker with direct patient contact.
* Have household contacts who are <2 years old or >80 years old or infirm or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease)
* Pregnancy, risk of pregnancy, or lactation (female subjects only).
* Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
* Regular use of laxatives, antacids, or other agents to lower stomach acidity.
* Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period. (Topical and intra-articular steroids will not exclude subjects).
* Known allergy to quinolones, trimethoprim-sulfamethoxazole or penicillins.
* Symptoms consistent with Traveller's Diarrhea concurrent with travel to countries where ETEC infection in endemic (most of the developing world) within 2 years prior to vaccination.
* Received vaccination against, or ingestion of, ETEC, cholera toxin, or LT toxin within 3 years prior to vaccination.
* Use of antibiotics during the 7 days prior to vaccination and/or proton pump inhibitors, H2 blockers, or antacids within 48 hours prior to vaccination.
* History of diarrhea in the 7 days prior to vaccination (outpatient diarrhea is defined as ≥ 3 unformed loose stools in 24 hours).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events and determination of systemic immune response and mucosal immune response | 13 weeks

SECONDARY OUTCOMES:
Assessing intestinal colonization by the vaccine ACE527 | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Harro, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research CIR, Baltimore, Maryland, United States